CLINICAL TRIAL: NCT07244744
Title: Investigating the Mechanisms of Short- and Long-term Responses to IL-23 Inhibition Using Tildrakizumab in Moderate to Severe Plaque Psoriasis Using High-definition Multiomics
Brief Title: Tilrdakizumab Almirall
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Other Study IDs: Tilrdakizumab Almirall
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — tildrakizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Biological: Tildrakizumab — Tildrakizumab, a monoclonal antibody targeting IL-23 p19, reduces inflammation in moderate to severe plaque psoriasis. Administered subcutaneously it improves skin symptoms and is well tolerated.

SUMMARY:
Define the mechanisms underlying the short- and the long-lasting effects of IL-23 targeting in plaque PsO, by characterizing the longitudinal effects of IL-23 inhibition on the ratio of Trm/Treg cells in the skin of moderate to severe plaque PsO patients. HDST (Visium HD) and HDSP (MICS) are used to characterize the early (2 weeks) and late (16 weeks) molecular effects of treatment with tildrakizumab on the skin of three patients with moderate to severe plaque psoriasis. Non-lesional and lesional skin samples taken at the start of treatment with tildrakizumab will be used, as well as healed skin adjacent to the original sampling sites at week 2 and week 16 after the start of treatment with tildrakizumab. The same samples will be examined using Visium HD and the MACSima imaging system.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older) with a diagnosis of moderate to severe chronic plaque psoriasis.
* Patients eligible for treatment with an IL-23 inhibitor, specifically Tildrakizumab.

Exclusion Criteria:

* Patients unable to comply with the study requirements.
* Known hypersensitivity to IL-23 inhibitors.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (18 years and older) with moderate to severe plaque psoriasis. These patients have a confirmed diagnosis and are eligible for treatment with Tildrakizumab. These patients are selected from existing biobank samples with informed consent for molecular analysis related to IL-23 inhibition.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in tissue-resident memory T cells (Trm) to regulatory T cells (Treg) ratio in lesional, non-lesional, and resolved skin at weeks 2 and 16 after Tildrakizumab treatment, assessed by high-definition spatial transcriptomics (Visium HD) and high-dimen | Assessment of changes in Trm/Treg cell ratio at early (2 weeks) and late (16 weeks) time points after initiation of Tildrakizumab treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CCIM, Institut für Entzündungsmedizin UKSH Lübeck, Lübeck, <Keine Auswahl>, Germany

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-10-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT07244744/Prot_000.pdf